CLINICAL TRIAL: NCT03918746
Title: The Feasibility of the Internet Attachment-Based Compassion Therapy (iABCT) for General Population
Brief Title: Feasibility of the Internet Attachment-Based Compassion Therapy (iABCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Collaborators: Generalitat Valenciana (Other); European Social Fund (Other)
Responsible Party: Principal Investigator, Daniel Campos Bacas, Principal Investigator, Universitat Jaume I
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UJaumeICO_CD/005/2019
Record Dates: First submitted 2019-04-11; First posted 2019-04-17 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Mental Health Wellness 1; Compassion
Keywords: compassion; internet-based Interventions; feasibility; meditation; attachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- internet Attachment-Based Compassion Therapy (iABCT) (Experimental): The intervention will consist of an internet version of Attachment-Based Compassion Therapy (iABCT).
  The length of the intervention will depend on the pace of each participant that will be advised to carry out one module per week, taking days between sessions to complete homework assignments. It is estimated that the online intervention can be completed in eight weeks, with a maximum period of ten weeks. However, each participant will be free to advance at his/her own pace. Formal telephone support will be not systematically provided, but participants will contact for technical assistance (i.e., web accessibility problems or forgotten password) if necessary.
  Interventions: Behavioral: internet Attachment-Based Compassion Therapy (iABCT)

INTERVENTIONS:
Behavioral: internet Attachment-Based Compassion Therapy (iABCT) — The internet version of Attachment-Based Compassion Therapy (iABCT) will be developed to be totally self-applied over the Internet through the website www.psicologiaytecnologia.com designed by Labpsitec (Laboratory of Psychology and Technology, Universitat Jaume I, and University of Valencia). The iABCT will consist of eight sequential modules: Module 0) Welcome module: approaching to the compassion; Module 1) Preparing ourselves for compassion. Kind attention; Module 2) Discovering our compassionate world; Module 3) Developing our compassionate world; Module 4) Understanding our relationship with compassion; Module 5) Working on ourselves; Module 6) Understanding the importance of forgiveness; Module 7) Consolidating the practice of compassion
  The content will present through texts, audios, videos, pictures, vignettes, and interactive exercises. Downloadable PDF files will be available so that users can review them offline.

SUMMARY:
The purpose of this study is to investigate the feasibility, acceptability and preliminary efficacy of the internet Attachment-based compassion Therapy (iABCT) to promote wellbeing and mental health for the general population.

A feasibility open trial and single-arm study will be conducted with three measurement points: at baseline (pre-intervention), immediately after the intervention (post-), and 3-month follow-up, where participants will be allocated to iABCT.

To the best of our knowledge, this is the first study to explore the feasibility and preliminary efficacy of Compassion-based Intervention (CBI) delivered over the internet in Spanish.

DETAILED DESCRIPTION:
Compassion refers to a multidimensional psychological construct that involves the feeling that arises in presence of another's suffering and implies the desire to help. There is a growing number of studies pointing out the benefits of Compassion-based Interventions (CBI) and their association with psychological health. CBI are focused on training compassion to others and/or towards oneself (self-compassion) employing formal and informal meditation practices. Recent scientific literature is emerging to prove the feasibility and efficacy of cultivating compassion over the Internet and, thus, delivering self-applied online CBI.

The aim of this study is to investigate the feasibility and acceptability of the internet Attachment-based compassion Therapy (iABCT) to promote wellbeing and mental health for the general population. A secondary aim is to explore the preliminary efficacy of iABCT at post-intervention and 3-month follow-up.

The principal hypothesis is that the iABCT will be feasible and well-accepted by participants in terms of expectations, satisfaction, usability, opinion, and cost-effectiveness. Moreover, it is expected that the iABCT will be effective to promote changes in self-reported measures of compassion, self-compassion, mindfulness, self-criticizing, attachment, wellbeing, and mental health. It is also hypothesized that gains will be maintained at 3-month follow-up.

A minimum of 35 participants is considered enough to cover the aims of this feasibility study and to provide precise and efficient estimations of parameters (i.e., means, standard deviations, effect size, and confidence intervals) for powering a larger randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years old or over.
* Have adequate knowledge to understand and read Spanish.
* Have a computer with speakers and Internet access in a secure setting (home or private office).
* Have an email account.
* Ability to use a computer and to surf the Internet.

Exclusion Criteria:

* Diagnosis of mental disorder according to the Diagnostic and Statistical Manual for Mental Health Disorders-Version 5 (DSM-5).
* Abuse or dependence on alcohol or other substances.
* Be receiving psychiatric or psychological treatment,
* Be engaged in ongoing formal meditation training (e.g., mindfulness or compassion intervention).
* Presence of heart disease, cardiorespiratory illness, or other severe medical condition.
* History of epileptic crisis.
* Unavailability to complete the online intervention because of operation or medical intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Changes in Pemberton Happiness Index (PHI) (Hervás & Vázquez, 201) | Before the intervention, immediately after the intervention, and 3-month follow-up after the intervention
  PHI is a measure of well-being that contains 11 items (in a scale from 0 to 10 point) related to different domains of remembered wellbeing, and 10 items related to experienced well-being (i.e., 5 positive and 5 negative emotional events that might have happened the day before) (answering YES/NO). The sum of these items produces a combined well-being index ranging from 0 to 10. Higher values represent higher wellbeing.

SECONDARY OUTCOMES:
Changes in Self-Compassion Scale (SCS-26) (Neff, 2003; García-Campayo et al., 2014) | Before the intervention, immediately after the intervention, and 3-month follow-up after the intervention
  The Self-Compassion Scale (SCS-26) is a 26-item questionnaire designed to assess overall self-compassion (total score) and three self-compassion facets: self-kindness (SCS-SK), common humanity (SCS-CH) and mindfulness (SCS-M). The Spanish version of the SCS-26 has shown high internal consistency and high test-retest reliability. The items are rated on a five-point Likert scale with 1 indicating almost never and 5 indicating almost always. After reversing the negatively formulated items, higher scores indicate greater self-compassion.
Changes in Compassion Scale (Pommier, 2000) | Before the intervention, immediately after the intervention, and 3-month follow-up after the intervention
  The Compassion Scale assesses compassion for others in similar dimensions to self-compassion. Responses are given on a 5-point scale ranging from 1 (almost never) to 5 (almost always). Pommier's (2010) results suggest that this scale presents good internal consistency and adequate convergent validity. A Spanish adaptation of Pommier's scale was developed for Brito-Pons (2014). The English version was translated by the researcher and refined with a team of psychologists and mindfulness instructors following a committee approach (Graham et al. 2003); finally, it was back-translated by native English speakers. Higher scores indicate greater compassion.
Changes in Forms of Self-Criticizing/Attacking and Self-Reassuring Scale-Short form (FSCRS-SF) (Sommers-Spijkerman et al., 2017) | Before the intervention, immediately after the intervention, and 3-month follow-up after the intervention
  The FSCRS-SF contains 14 items to assesses two forms of self-criticism: inadequate self and hated self, and the ability to self-reassure.
  Participants respond to a selection of statements, asking about how one thinks and reacts in the face of failures or setbacks, on a 5-point Likert scale ranging from 0 (not like me at all) to 4 (extremely like me). Higher scores indicate a greater sense of inadequacy, self-hate, or self-reassurance. The FSCRS-SF subscale scores had adequate test-retest reliability and satisfactory convergent validity estimates with theoretically related constructs.
Changes in Five Facets of Mindfulness Questionnaire (FFMQ-15) | Before the intervention, immediately after the intervention, and 3-month follow-up after the intervention
  The FFMQ-15 is a short version of the FFMQ-39. This version includes 15 items to assess dispositional mindfulness rated on a Likert scale ranging from 1 (never or very rarely true) to 5 (very often or always true).
  Five facets of mindfulness are assessed: Observe, refers to the subject's capacity to pay attention to internal and external experiences such as sensations, thoughts, or emotions; Describe, measures the ability to describe events and personal responses in words; Acting with awareness, includes focusing on the activity being carried out, as opposed to behaving automatically; Non-judging of inner experience, refers to the ability to take a non-evaluative stance toward thoughts and feelings; and Non-reactivity to inner experience, allowing thoughts and feelings to come and go, without getting caught up in them or carried away by them. The five scales show good internal consistency. Higher scores represent higher compassion.
Changes in Relationships Questionnaire (RQ) (Bartholomew y Horowitz, 1991; Alonso-Arbiol y S.Yárnoz-Yaben, 2000). | Before the intervention, immediately after the intervention, and 3-month follow-up after the intervention
  The RQ uses a 7-point Likert-scale that assesses and matches participants with one of four attachment styles: (i) secure, (ii) pre-occupied, (iii) dismissive and (iv) fearful. A mathematical calculation permits a categorical assessment of attachment style (i.e. secure or insecure) (Griffin & Bartholomew 1994), and qualitative self-descriptor criteria can be used for confirmatory purposes. Studies have demonstrated that the reliability of the self-descriptor criteria is high (Leak and Parsons 2001; Yarnoz-Yaben and Comino 2011). The RQ also offers the possibility of measuring two key dimensions underlying attachment in adults (Griffin and Bartholomew 1994a)-namely, anxiety, which relates more to the self, and avoidance, which relates more to others (Griffin and Bartholomew 1994b). The anxiety dimension is calculated using the sum of the four attachment style ratings. High scores in this dimension reflect high anxiety towards social relationships.
Changes in General Health Questionnaire (GHQ-12) (Rocha et al., 2011) | Before the intervention, immediately after the intervention, and 3-month follow-up after the intervention
  GHQ-12 is one of the most widely used screening tests to assess mental health of a population, and is designed as a structured, brief and self-administered questionnaire.
  Every one of its 12 items regarding recent symptoms, feelings or behaviors is answered on a four-category Likert scale. Categories 1 and 2 are given value 0, and categories 3 and 4 are given value 1. Values from 12 items are added together to get an overall score. A probable psychiatric case is considered when the score is equal to or greater than 3.
Changes in Non-Attachment Scale (NAS-7) (Feliu et al., 2016; Sahdra et al. 2015) | Before the intervention, immediately after the intervention, and 3-month follow-up after the intervention
  The NAS-7 is scored on a 6-point scale ranging from 1 = disagree strongly to 6 = agree strongly and designed to measure nonattachment (e.g., I can let go of regrets and feelings of dissatisfaction about the past when pleasant experiences end, I am fine moving on to what comes next).
  The NAS-7 is unifactorial and shows excellent internal consistency (α = .82).
  Higher scores represent higher nonattachment values.
Changes in International Positive and Negative Affect Schedule Short Form (I-PANAS-SF; Thompson, 2007) | Before the intervention, during the intervention, immediately after the intervention, and 3-month follow-up after the intervention
  The I-PANAS-SF -a reduced version of the PANAS- is composed of 10 items with 5-item Positive Affect (PA) Negative Affect (NA) subscales.
  In a series of validation studies (N = 1,789), the cross-sample stability, internal reliability, temporal stability, cross-cultural factorial invariance, and convergent and criterion-related validities of the I-PANAS-SF were examined and found to be psychometrically acceptable.
  Higher scores of PA subscale represent higher positive affect. Higher scores of NA subscale represent higher negative affect.
Changes in Purpose-In-Life Test (PIL-10) (García-Alandete, Rosa, y Sellés, 2013; García-Galante, 2014) | Before the intervention, immediately after the intervention, and 3-month follow-up after the intervention
  The PIL test is a 10-item self-report attitudinal scale designed to measure the extent to which a respondent perceives a general sense of meaning and purpose in life or respectively suffers from an "existential vacuum". The Spanish validation has shown to be a reliable measure to assess the meaning of life. Higher scores represent a higher sense of meaning and purpose in life.
Changes in Compassion Practice Quality Questionnaire(12 ítems) (adapted from Del Re et al., 2015). | During the intervention, immediately after the intervention, and 3-month follow-up after the intervention
  The Compassion Practice Quality Questionnaire has been developed for this study to assess difficulties related to the practice of compassion meditation. This self-reported questionnaire includes 10 items that participant scores on a scale ranging from 0 to 100 indicating the percentage of time that his/her experience reflects each statement. Higher scores represent higher difficulties related to the compassion meditation practice.

OTHER OUTCOMES:
Attrition rate | Immediately after the intervention, and 3-month follow-up after the intervention
  Percentage of participants that drop-out the intervention after having access for first time. Higher scores represent higher drop-out rates.
Expectations and satisfaction Questionnaire (Adapted from Borkovec y Nau, 1972) | Before the intervention, immediately after the intervention, and 3-month follow-up after the intervention
  These questionnaires were adapted from Borkovec and Nau (1972) to measure participant expectations before the intervention and their later satisfaction with it.
  Each scale includes six items rated from 0 ("not at all") to 10 ("very much"). The questions addressed how logical the intervention seemed, to what extent the participant expected to be satisfied with it, whether the participant would recommend the intervention to others, whether it would be useful for psychological problems, the interventions' usefulness for the participants, and to what extent it could be aversive (reverse item). Higher scores represent higher expectations and satisfaction levels.
Acceptability and Usability Questionnaire (Labpsitec, 2019) | immediately after the intervention, and 3-month follow-up after the intervention
  This instrument was adapted from the System Usability Scale (SUS) in order to assess the usability of a service or product and the acceptance of technology by the people who use it. The SUS has been shown to be a valuable and robust tool for assessing the quality of a wide range of user interfaces, as it is easy to use and understand. This scale includes 10 statements rated on a five-point scale measuring agreement with the statement (0 = strongly disagree; 4 = strongly agree). The final score is obtained by adding the scores on each item and multiplying the result by 2.5. Scores range from 0 to 100, where higher scores indicate better usability.
Qualitative opinion interview | immediately after the intervention
  Qualitative Interview has been specifically developed to assess participant opinions about the internet intervention. This interview included 14 questions: seven of them regarding usefulness of the intervention, components, modules, information provided, and multimedia elements (e.g., images, audios, videos, pdf) rated on a scale from 1 to 5 (1 = very little; 2 = little; 3 = something; 4 = a lot; and 5 = very much) and two dichotomous questions ("yes" or "no") regarding whether they would like having at their disposal the program for more time after the treatment has finished, as well as whether they would like to have longer access. Additionally, options to extend the participants' qualitative responses were available. Finally, two open questions are included to assess advers or unwanted effects and facilitators and barriers towards the intervention received.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Campos, PhD, Principal Investigator — Universitat Jaume I. Instituto de Investigación Sanitaria Aragón (IIS Aragón).
Locations (1):
- Centro de Salud Arrabal, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
The raw IPD will be made available by the authors, without undue reservation, to any qualified researcher. Dataset will be available through scientific repositories and via email request.
Supporting Information: Study Protocol, SAP
Time Frame: When the study is finished and results published.
Access Criteria: The raw IPD will be made available by the authors, without undue reservation, to any qualified researcher.

REFERENCES:
- [Background] García-Campayo J, Demarzo M. Mindfulness y compasión. La nueva revolución. Barcelona: Siglantana; 2015.
- [Background] García-Campayo J, Navarro-Gil M, Demarzo M. Attachment-based compassion therapy. Mindfulness & Compassion. 2016;1:68-74. doi:10.1016/j.mincom.2016.10.004.
- [Background] Effects of Attachment-Based Compassion Therapy (ABCT) on Self-compassion and Attachment Style in Healthy People. Mindfulness
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. Pilot Feasibility Stud. 2016 Oct 21;2:64. doi: 10.1186/s40814-016-0105-8. eCollection 2016. PMID 27965879
- [Background] Krieger T, Martig DS, van den Brink E, Berger T. Working on self-compassion online: A proof of concept and feasibility study. Internet Interv. 2016 Oct 8;6:64-70. doi: 10.1016/j.invent.2016.10.001. eCollection 2016 Nov. PMID 30135815
- [Derived] Campos D, Navarro-Gil M, Herrera-Mercadal P, Martinez-Garcia L, Cebolla A, Borao L, Lopez-Del-Hoyo Y, Castilla D, Del Rio E, Garcia-Campayo J, Quero S. Feasibility of the Internet Attachment-Based Compassion Therapy in the General Population: Protocol for an Open-Label Uncontrolled Pilot Trial. JMIR Res Protoc. 2020 Aug 14;9(8):e16717. doi: 10.2196/16717. PMID 32384051
- See also: Psychology and Technology website — https://www.psicologiaytecnologia.com/